CLINICAL TRIAL: NCT06534164
Title: Telerehabilitation of Balance Clinical and Economic Decision Support System
Acronym: TeleRehab DSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National and Kapodistrian University of Athens (Other); University Medical Center Freiburg (Other); King Chulalongkorn Memorial Hospital (Other); Secretaria Regional de Saúde e Proteção Civil da Região Autónoma da Madeira (Unknown); Institute of Communications and Computer Systems, Athens, Greece (Other); University of Ioannina (Other); Vilabs (Unknown); BioIRC (Unknown); Activage (Unknown); Institue De Desenvolvimento De Novas Technologiassociacao (Unknown); Quantitas SRL (Unknown); Instituto para o Desenvolvimento e Inovação (Unknown); BRIDG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCLondon 101057747; 101057747 (Other Grant/Funding Number: European Union Horizon Europe)
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Mild Cognitive Impairment; Vestibular Diseases; Long Covid19
Keywords: vestibular; rehabilitation; falls; balance; exercise; artificial intelligence; telerehabilitation; physiotherapy; cognitive
MeSH Terms: conditions — Stroke; Cognitive Dysfunction; Vestibular Diseases; Post-Acute COVID-19 Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is an assessor-blinded, parallel, randomised controlled study. Participants will be block randomised by condition (stroke, MCI, long covid-19, vestibular disorders) using an online platform into either the intervention group (IG) or control group (CG). Within the IG, participants will be randomised into one of two groups; 1) High tech TeleRehab DSS system, 2) Low tech TeleRehab DSS system. Participants will not be able to choose their preferred group and must be willing to participate in the assigned group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors will be blinded to which study arm participants have been allocated to. Due to the nature of the study, investigator's and participants cannot be blinded, althouhg intervention group participants will be blinded as to which intervention (High vs. Low tech) they have been allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Full/High-tech TeleRehab DSS (Experimental): 5x/week x 9 weeks All TeleRehab DSS components: multisensory balance exercises, AR avatar, real-time feedback, AR gamified activities, sensor-monitored exercise performance and additional cognitive training.
  Interventions: Device: Full/High Tech Telerehabilitation decision support system
- Basic/Low-tech TeleRehab DSS (Experimental): 5x/week x 9 weeks With depth camera, motion sensors and tablet for multisensory balance exercises, real time feedback, sensor monitored exercise performance and cognitive games.
  No exergames, no smartwatch, no mobile phone.
  Interventions: Device: Basic/Low Tech Telerehabilitation decision support system
- OTAGO Home Exercise programme (Active Comparator): 9-week balance exercise programme developed by a research group at University of Otago, New Zealand [12]. The OTAGO HEP will be provided to all individuals in the control arm who report falls/are at risk of falls. The OTAGO group participants will receive a pamphlet with instructions for home exercises within the programme, resistance bands and an exercise diary.
  The OTAGO HEP booklet is available at https://www.livestronger.org.nz/assets/Uploads/acc1162-otago-exercise-manual.pdf
  Interventions: Procedure: OTAGO Home exercise program
- Vestibular rehabilitation programme (Active Comparator): Daily x 9 weeks For participants with problems chronic (lasting >3 months) dizziness/imbalance due to chronic vestibular disorder (affecting the vestibular /balance system) or due to long Covid). The vestibular rehabilitation group participants will receive a booklet with vestibular exercises which have been individualised based on the assessment by the research team member. The exercise booklet is a validated and widely used intervention for vestibular disorder [17]. This will be provided to all individuals in the control arm with chronic dizziness/imbalance (>3 months) without falls/risk of falls (FGA>22).
  The booklet has descriptions and diagrams of the exercises and instructions on how to progress these as well as an exercise log, available at: https://www.menieres.org.uk/files/pdfs/balance-retraining-2012.pdf
  Interventions: Procedure: Vestibular rehabilitation program

INTERVENTIONS:
Device: Full/High Tech Telerehabilitation decision support system — The TeleRehaB DSS intervention includes balance rehabilitation programme delivered via an augmented reality hologram of a virtual physiotherapist. The system delivers exercises demonstrated via a hologram of the physiotherapist and corrected in real time by the hologram prompts based on performance monitoring via sensors. It includes different multisensory balance and gait exercises, physical activity and memory training and exergames (video games which are also exercises) to improve balance function in older adults. The system can thus assess and remotely monitor how users are performing the exercises.
  Exercise progressions will be suggested by the AI-supported TeleRehaB DSS and approved by the clinicians, which will be loaded into the participant's programme.
  Arms: Full/High-tech TeleRehab DSS
Device: Basic/Low Tech Telerehabilitation decision support system — The basic system does not inlcude exergames, a smartwatch, or a mobile phone for activity tracking.
  It includes different multisensory balance and gait exercise, cognitive training and real-time feedback from motion sensors.
  Exercise progressions will be suggested by the AI-supported TeleRehaB DSS and approved by the clinicians, which will be loaded into the participant's programme.
  Arms: Basic/Low-tech TeleRehab DSS
Procedure: OTAGO Home exercise program — balance rehabilitation program
  Arms: OTAGO Home Exercise programme
Procedure: Vestibular rehabilitation program — vestibular rehabilitation and dizziness program
  Other Names: Meniere's Dizziness Booklet
  Arms: Vestibular rehabilitation programme

SUMMARY:
This study follows the successfully completed HOLOBalance project which was funded by the EU Horizon 2020 scheme. TheHOLOBalance platform delivers exercises demonstrated via a hologram of the physiotherapist and corrected in real time by the hologram prompts based on performance monitoring via sensors. Further information is available at: https://holobalance.eu/. HOLOBalance was developed as a comprehensive rehabilitation protocol for individualised remote (tele)rehabilitation balance physiotherapy programme. It includes different multisensory balance and gait exercises, physical activity and memory training and exergames (video games which are also exercises) to improve balance function in older adults. The system can thus assess and remotely monitor how users are performing the exercises.

This multisite randomised control trial (TeleRehab DSS, short for TeleRehabilitation Decision Support System) aims to (i) determine the system's safety, acceptability, and feasibility explore effectiveness of running such programme in comparison with the current standard care for middle-age/older adults with balance disorders/falls due to MCI, vestibular disorders, stroke or long Covid. This study also aims to (ii) assess if balance function, gait, cognitive function, balance confidence, and wellbeing can improve more compared to standard intervention and (iii) provide preliminary data for a definitive randomised controlled trial.

This study involves human participants, and each clinical site has applied for appropriate ethical approval.

DETAILED DESCRIPTION:
This is an assessor-blinded (researchers assessing the participants will not know what study group participants will be in), randomised (participants will join different study groups randomly) controlled study. Participants will be randomised using an online platform to undergo a home-based exercise programmes, into either the intervention group (IG) or control group (CG). Participants will not be able to choose their preferred group and must be willing to participate in the assigned group.

All study participants will attend two sessions at UCL. The first assessment will be within one week prior to starting the programme, and the second will be within one week of completing the programme. Participants will be asked to complete a questionnaire set, walking/balance tests and a cognitive test.

Participants will receive telephone calls each week to monitor their progress. Participants will also receive remote program reviews at weeks 3, 6 and 9, from a member of the research team to assess and change exercises as required. Participants will be advised to contact the research team by email or by telephone during working hours if they have concerns or questions about their rehabilitation program or the TeleRehab DSS system. The research team will judge whether an additional home visit is required. If a patient does not complete their exercises for three consecutive days, a flag/warning will appear on the patients dashboard as a priority patient to follow up with, within 24 hours.

Intervention Group (IG): TeleRehab DSS The intervention (TeleRehaB DSS) group participants will be visited by a research team member to install the TeleRehab DSS system in their home and taught how to use the system, with a practice session. The system comprises a depth camera, lightweight augmented reality headset that displays the hologram, body-worn sensors that record movements and a heart rate sensor. Participants will be required to wear all the equipment when performing the prescribed exercises. A demo-video (including equipment and hologram) is available at www.holobalance.eu. Exercise progressions will be suggested by the AI-supported TeleRehaB DSS and approved by the clinicians at weeks 3, 6, and 9, which will be loaded into the participant's programme. At the end of the study, participants will be invited to take part in an interview to discuss their experience with using the TeleRehab DSS system.

The IG will receive the TeleRehaB DSS supported, prescribed, progressed and delivered intervention. In the TeleRehaB DSS IG, the platform will suggest two possible management strategies, on an individualized basis, based on patient profiles and expected benefit: 1)The high-tech, full TeleRehaB DSS with all components of the intervention consisting of TeleRehaB DSS AI-progressed multisensory balance exercises with the use of the AR avatar, real time feedback, AR gamified intervention, sensor monitored exercise performance and additional cognitive training, 2) the low-tech, basic version of TeleRehaB DSS, with depth camera, sensors and tablet - multisensory balance exercises, real time feedback, sensor monitored exercise performance and cognitive games, with no exergames, no smartwatch, and no mobile phone. The clinician can override the TeleRehab DSS group allocation decision if it is deemed unsafe. The intervention will be delivered as a daily (5 days per week, 12 weeks long) home-based exercise programme prescribed by non-experts (junior physiotherapist without vestibular expertise or non physio) with DSS support and coaching.

Control group (CG):

Control group participants will receive standard balance rehabilitation. Stroke and mild cognitive impairment (MCI) participants will receive the OTAGO home exercise program, while vestibular dysfunction and long covid-19 participants will receive the Meniere's Dizziness Booklet program.

1. OTAGO Home Exercise Programme (HEP), a balance exercise programme developed by a research group at University of Otago, New Zealand. The OTAGO HEP will be provided to all individuals in the control arm who report falls/are at risk of falls. The OTAGO group participants will receive a pamphlet with instructions for home exercises within the programme, resistance bands and an exercise diary. The OTAGO HEP booklet is available at https://www.livestronger.org.nz/assets/Uploads/acc1162-otago-exercise-manual.pdf
2. Vestibular rehabilitation programme - for participants with problems chronic (lasting >3 months) dizziness/imbalance due to chronic vestibular disorder (affecting the vestibular /balance system) or due to long Covid). The vestibular rehabilitation group participants will receive a booklet with vestibular exercises which have been individualised based on the assessment by the research team member. The exercise booklet is a validated and widely used intervention for vestibular disorder. This will be provided to all individuals in the control arm with chronic dizziness/imbalance (>3 months) without falls/risk of falls (FGA>22). The booklet has descriptions and diagrams of the exercises and instructions on how to progress these as well as an exercise log, available at: https://www.menieres.org.uk/files/pdfs/balance-retraining-2012.pdf

ELIGIBILITY:
ALL PARTICIPANT Inclusion Criteria:

* Age 40-80 years
* community dwelling able to walk 500-m independently or with a stick
* Depression subscale on Hospital Anxiety and Depression Scale <10/21 (14-item questionnaire)
* No significant visual impairment (as self-reported by participants)
* Willing to comply with study procedures, proposed training and testing regime
* With capacity to consent
* No acute musculoskeletal or other injuries that would prevent participation in a structured exercise program
* Is not currently, and has not in the past 8-weeks received any falls/balance/vestibular and/or cognitive rehabilitation.
* Does not any implanted medical devices or a cardiac pacemaker.
* Does not have any other co-existing neurological conditions (ie. Multiple sclerosis, Parkinson's disease, neuropathy etc.)
* Does not have any language or communication deficits impairing their ability to communicate and/or express their thoughts.
* Has at least one functional hand for grip function and computer use.
* Fulfilling all of the criteria from one of the below sub-groups

STROKE COHORT who will fulfil the additional criteria:

* Individuals with diagnosis of focal ischaemic or haemorrhagic stroke, as confirmed by a clinical letter.
* Onset >/= 3 months prior to study.
* Montreal Cognitive Assessment (MoCA) score n >/=23
* At risk of falls (i.e. Functional Gait Assessment FGA score </=22/30; FGA is a validated quick balance task assessment) AND/OR having experienced a fall(s) in the last 12 months

MCI COHORT who will fulfil the additional criteria:

* Individuals with new or existing formal diagnosis of MCI, according to the International Classification of Disease 10 (ICD10) , as confirmed by a clinical letter.
* At risk of falls (FGA </= 22/30) AND/OR having experienced a fall(s) in the last 12 months.

VESTIBULAR COHORT who will fulfill the additional criteria

* Montreal Cognitive Assessment (MoCA) score n >/=23
* Individuals with a diagnosis of a vestibular disorder (peripheral and/or mixed peripheral and central):
* Peripheral vestibular disorder in which the balance problem lies in the vestibular/balance system within the inner ear.
* Mixed vestibular disorder in which the balance problem lies in the vestibular/balance system within the inner ear (peripheral) and involving the nerves or neuronal network in the brain/brainstem responsible for balance (central).
* Chronic dizziness and/or unsteadiness (>/= 3 months duration) that started at the time or after the vestibular disorder diagnosis.
* Dizziness handicap inventory (DHI >34) AND/OR At risk of falls (FGA </=22/30)

LONG COVID-19 COHORT who will fulfill the additional criteria:

* Montreal Cognitive Assessment (MoCA) score n >/=23
* Individuals with laboratory confirmed diagnosis of Covid (>/=6 months prior to study onset), as confirmed by a clinical letter.
* Who have been diagnosed with long Covid, as confirmed by a clinical letter.
* Who have chronic dizziness and/or unsteadiness which started after the Covid illness (self-report by the patient; duration </=3 months).
* Dizziness handicap inventory (DHI >34) AND/OR At risk of falls (FGA </=22/30)

Exclusion Criteria:

* Outside of the stated age bracket
* Unable to walk independently (even with use of a walking stick)
* MOCA score <23
* Score of 10 or higher on depression subscale of HADS
* Unwilling to comply with study procedures, proposed training and testing regime
* No capacity to consent
* Significant visual impairment or homonymous hemianopia (stroke cohort only) (self-reported)
* Orthostatic hypotension or uncontrolled hypertension
* Other neurological problem (e.g. Parkingson's disease, Multiple Sclerosis etc.)
* Language and communication deficits impairing ability to express thoughts (e.g. Aphasia)
* Has participated in a clinical drug trial in the past 6 months.
* Acute musculoskeletal injury that prevents participation in a structured exercise programme (e.g. lower limb fracture).
* Has an implanted medical device or cardiac pacemaker.
* Diagnosis of unstable Meniere's or with more than 4 migraines/month at the time of participating in the study
* Not fulfilling the inclusion criteria for one of the sub-groups (such as criteria for Stroke group, or MCI group, or chronic vestibular disorder group, or long-Covid group), as outlined above.
* Unable to provide a clinical letter confirming diagnosis.
* For those with stroke, no visual spatial neglect.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate (acceptability) | Baseline (week 0) through to post-intervention at week 10
  percentage of recruited participants that were eligible
Incidence of Treatment-Emergent Adverse Events (safety) | Baseline (week 0) through to post-intervention at week 10
  Participants will be monitored for adverse events during telephone or face-to-face contacts as part of the intervention phase and during follow-up assessments. Any adverse events related to the treatment will be reported via an adverse events form on the system database. Falls diaries will be collected weekly from participants during the intervention and monthly for up to 6 months after completion of the intervention.
Feasibility (protocol deviations/problems) | Baseline (Week 0) through to post-intervention at week 10
  Incidence of protocol deviation and/or implementation problems reported during the intervention.
Participants experience using the system (usability) | weekly and post-intervention at week 10
  Participants experience using the system (perceived benefits) via via weekly check in on frustration levels, technical troubleshooting and any other usability considerations, as well as during exit interviews for all TeleRehab DSS group completers.
Adherence to Intervention | Week 1 through to completion at week 9
  percentage of prescribed sessions completed throughout the intervention
Drop-out rate (acceptability) | Baseline (week 0) through to post-intervention at week 10
  Percentage of enrolled participants that were loss to follow-up or drop-outs

SECONDARY OUTCOMES:
Mini Balance Evaluation Systems Test (Mini-BESTest) | Baseline (week 0) & post intervention (Week 10)
  a 14-item test that assesses dynamic balance, on a scale of 0 (indicating severe balance impairment) to 28 (representing normal balance with a total score of 28 points.
Functional Gait Assessment (FGA) | Baseline (week 0) & post intervention (Week 10)
  test that assesses complex gait tasks (e.g. walking with head turns or stopping and turning, 5 minutes).
Incremental cost-effectiveness ratio (ICER) | 1 year before study to 1 year after the end of the intervention
  Cost-effectiveness, by dividing the difference in mean QALYs; The Incremental Cost-Effectiveness Ratio (ICER) is calculated as the difference in cost (ΔC) divided by the difference in effectiveness (ΔE) between two interventions. Lower ICER values indicate better cost-effectiveness, while higher values suggest greater cost per unit of effectiveness gained. An intervention is considered cost-effective if its ICER falls below a predefined willingness-to-pay (WTP) threshold
EuroQol five dimensional descriptive system (EQ-5D-5L) | Baseline (week 0) & post intervention (Week 10)
  Measure of quality-adjusted life years (QALYs). EQ-5D-5L is a standardized, valid and reliable simple, generic measure of health status for clinical and economic appraisal. The respondent is asked to rate their health status on these five dimensions from 1 to 5 respectively as no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS (Visual Analogue Scale) records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. The respondent is asked to mark an X on the scale to indicate "how your health is TODAY" with a higher score indicating better health-related quality of life .
Montreal Cognitive Assessment (MoCA) | Baseline (week 0) & post intervention (Week 10)
  includes sections on visuospatial/executive function, naming, attention, language, abstraction, memory and orientation to time and place (6 questions) with a scor range from 0-30, with a higher score indicating better cognitive function.
Rapid Assessment of Physical Activity (RAPA) | Baseline (week 0) & post-intervention (Week 10)
  The 9-item self-administered Rapid Assessment of Physical Activity (RAPA) is a questionnaire that assesses levels of a wide range of physical activity level in adults older than 50 years, with a score range 1-7 and a higher score indicating ihgher levels of physical activity.
Dizziness Handicap Inventory (DHI) | Baseline (week 0) & post intervention (Week 10)
  The 25-item self-report Dizziness Handicap inventory (DHI) validated questionnaire that assesses functional, emotional and physical domains. Responses are graded 0 (no), 2 (sometimes) or 4 (yes) with higher scores indicating greater impact of dizziness maximum and maximum score of 100 points (15 minutes).
The Activities-specific balance confidence scale (ABC) | Baseline (week 0) & post intervention (Week 10)
  The Activities-specific Balance Confidence Scale (ABC) that assesses patient's perceived confidence for 16-activities of daily living without losing balance .Score range from 0-100 with higher schore indicating greater balance confidence and scores ≤67/100% indicate increased falls risk.
The Hospital Anxiety and Depression Scale (HADS-d) depression subscale | Baseline (week 0) & post intervention (Week 10)
  a 14-item scale which assesses non-somatic anxiety (HAD-A) and depression (HAD-D) symptoms. Scores range from 0-21 for each subscale, with higher scores indicating worse outcomes (greater anxiety or depression).
Fatigue Severity Scale (FFS) | Baseline (week 0) & post intervention (Week 10)
  a 9-item instrument designed to assess fatigue as a symptom of a variety of different chronic conditions and disorders. The scale addresses fatigue's effects on daily functioning, querying its relationship to motivation, physical activity, work, family, and social life, and asking respondents to rate the ease with which they are fatigued and the degree to which the symptom poses a problem for them. Sca;e 9-63 with higher score indicating greater fatigue.
Warwick-Edingburgh Mental Wellbeing Scale (WEMWBS) | Baseline (week 0) & post intervention (Week 10)
  developed to enable the measuring of mental wellbeing in the general population and the evaluation of projects, programmes and policies which aim to improve mental wellbeing. The 14-item scale WEMWBS has 5 response categories, summed to provide a single score. The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing, thereby making the concept more accessible. The scale has been widely used nationally and internationally for monitoring, evaluating projects and programmes and investigating the determinants of mental wellbeing. Scale 14-70 with higher score indicating better mental wellbeing.
Situational Vertigo Questionnaire(SVQ): | Baseline (week 0) & post intervention (Week 10)
  The SVQ is 20-item questionnaire designed to assess discomfort in situations of intense visual salience of visual-vestibular conflict. It was originally developed as a measure of space and motion discomfort. The questions are graded on a scale from 0 (not at all) to 4 (very much), with a higher score indicating greater vertigo severity.
The system Usability Scale (SUS) | post-intervention (week 10)
  The System Usability Scale (SUS) scale 1-5 rated on 10 aspects, with a total possible score of 0-100, with a higher score indicated better usability.
User experience questionnaire (UEQ) | Baseline (week 0), Week 8 & post intervention (Week 10)
  The User Experience Questionnaire (UEQ; scale 1-7 on 26 dimensions of attractiveness, perspicuity, efficiency, dependability, stimulation and novelty with a score range of -3 (worst) to +3 (best) with a higher score indicating a more positive user experience.
Falls | collected weekly for the duration of the 9-week intervention and up to 6 months after completing the intervention
  Falls diary collected (self-reported)
System performance | post-intervention (week 10)
  We will also compare the TeleRehaB DSS predicted versus observed patient outcomes on the EQ-5D-5L, and secondary outcome measures, to assess the system performance
eHealth Literacy Assessment (eHEALS) | Baseline (week 0)
  a 10-item likert scale questionnaire that evaluate's patients' skills in finding, evaluating and applying electronic health information. Responses range from 1 (strongly disagree, to 65 (strong agree), with total scores indicating levels of eHealth literacy. This will be used to help validate the AI-model in terms of participant allocation into the high-tech versus low-tech solution.
The Senior technology acceptance & adoption model (STAM) | Baseline (week 0)
  is a 38-item questionnaire, with items rated on a 1-10 Likert scale to measure factors influencing technology acceptance among older adults, with a higher scores indicating greater perceived digital literacy.
Mobile Device Proficiency Questionnaire - short (MDPQ-s) | Baseline (week 0)
  is a 16-question version of the full MDPQ-16. The MDPQ, its subscales, and the MDPQ-16 were found to be highly reliable and valid measures of mobile device proficiency in a large sample. We conclude that the MDPQ and MDPQ-16 may serve as useful tools for facilitating mobile device training of older adults and measuring mobile device proficiency for research purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Doris-Eva Bamiou, PhD, Principal Investigator — University College, London
Locations (5):
- University Medical Center Freiberg Neurocenter (UKLFR), Freiberg, Germany
- National and Kapodistrian University of Athens, Athens, Greece
- Secretaria Regional de Saúde e Proteção Civil da Região Autónoma da Madeira, Madeirã, Portugal
- King Chulalongeorn Memorial Hospital (KMCH), Bangkok, Thailand
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data collected willl be analysed, and a Final Study Report prepared. with results published in academic journals and disseminated in relevant clinical/scientific peer-reviewed literature and conferences. No participant identifiable data will be included in the final study reports or in the process of dissemination of the study results. The participants will be guided to where they can access the final result publication(s). The study protocol and study report will be published. Anonymised data will be uploaded to the Zenodo data repository and will be available to other researchers in line with open science principles. The research data collected in the course of the study will be retained by UCL and other clinical partners in their capacity as a sponsor for 20 years after the research study has ended. The data will be then securely destroyed.
Supporting Information: Study Protocol, ICF
Time Frame: 20 years after the research study has ended; Nov 2025 - Nov 2045
Access Criteria: All study research team members at all clinical sites will comply with their local requirements with regards to the collection, storage, processing and disclosure of personal information and will uphold the Act's core principles.
  The creation of coded, depersonalised data where the participant's identifying information will be replaced by an unrelated sequence of characters will be in place. The digital data collected will be stored in digital format at each clinical sites secure safe haven data platform with encrypted and password protection. The data (hard copies) collected during the study will be stored in the study site file in a securely locked designated cabinet at each clinical site for the duration of the study.

REFERENCES:
- See also: EQ-5D-5L — https://euroqol.org/information-and-support/euroqol-instruments/eq-5d-5l/
- See also: Functional Gait Assessment — http://geriatrictoolkit.missouri.edu/FGA/Wrisley-2007-FGA_PTJ_84-10-Appendix.pdf
- See also: mini Balance Evaluation Systems Test — http://www.bestest.us/files/7413/6380/7277/MiniBEST_revised_final_3_8_13.pdf
- See also: Montreal Cognitive Assessment (MoCA) — https://mocacognition.com/paper/
- See also: TeleRehab Website — http://telerehab-project.eu/
- See also: Rapid Assessment of Physical Activity — http://depts.washington.edu/hprc/programs-tools/tools-guides/rapa/
- See also: Dizziness Handicap Inventory — https://geriatrictoolkit.missouri.edu/vest/Dizziness-Handicap-Inventory.pdf
- See also: Activities Specific Balance Confidence Scale — https://sites.temple.edu/rtassessment/files/2018/10/Activities-Specific-Balance-Confidence-ABC-Scale.pdf
- See also: Hospital Anxiety and Depression Scale — https://www.svri.org/sites/default/files/attachments/2016-01-13/HADS.pdf
- See also: Fatigue Severity Scale — https://www.sralab.org/sites/default/files/2017-06/sleep-Fatigue-Severity-Scale.pdf
- See also: Warwick Edingburgh Mental Wellbeing Scale — https://warwick.ac.uk/fac/sci/med/research/platform/wemwbs/using/howto/
- See also: Situational Characteristics Questionnaire (SCQ) — https://neuropt.org/docs/vestibular-sig/situational_vertigo_questionnaireA068B2C6D4D5.pdf?sfvrsn=ef974640_4
- See also: System Usability Scale — https://www.usability.gov/how-to-and-tools/methods/system-usability-scale.html
- See also: User Experience Questionnaire — https://www.ueq-online.org/